CLINICAL TRIAL: NCT05281926
Title: A Phase I, Open-label Study to Assess the Safety and Efficacy of Poly-ICLC Plus Nivolumab in Unresectable Hepatocellular Carcinoma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 202104104MIND
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — poly ICLC; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Poly-ICLC (Experimental): Hiltonol is a poly-ICLC developed by the Oncovir, Inc. A phase I study of hiltonol monotherapy in solid tumors was completed (NCT01984892). Clinical trials of hiltonol plus ICIs are undergone in various type cancers (NCT03721679, NCT02834052).
  Interventions: Drug: Poly ICLC

INTERVENTIONS:
Drug: Poly ICLC — IT Poly-ICLC injection (1.0 mg) at Day 1 of weeks 0, 1 and 2. IM Poly-ICLC (20 μg/Kg) at Day 1 and Day 3 of weeks 3, 4, 5 and 6.
  Other Names: Nivolumab

SUMMARY:
Hepatocellular carcinoma (HCC) is a prevalent malignancy with great disease burden both in Taiwan and worldwide 1. Early stage HCC can be treated by surgical resection, radiofrequency ablation, embolization and liver transplantation. However, treatments for advanced HCC are still unsatisfactory. Systemic therapy is necessary for advanced HCC 2. Target therapy using sorafenib was established a decade ago, but its response rate is quite low (~3%), the adverse effects may be intolerable and it can only extend survival 2.3 to 2.8 months 3,4. Newly developed tyrosine kinase inhibitors (TKIs) include regorafenib 5, lenvatinib 6, cabozantinib 7 and ramucirumab 8. The single target therapy objective response rate is around 3-24%. Recently, immune checkpoint inhibitors (ICIs) emerged as a new hope for cancer therapy in various kinds of malignancies including HCC. These include CTLA4, PD-1 and PD-L1 blockades.

DETAILED DESCRIPTION:
This is an open-label, phase I pilot study. A total of 10 patients will be recruited in National Taiwan University Hospital between October, 01, 2021 and December, 31 2023. All examinations and treatment will be performed at National Taiwan University Hospital. The inclusion criteria are Child-Pugh classification A, unresectable HCC patients with age more than 20 years-old and radiologically measurable disease that is at least 2 cm in longest dimension of the target tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of hepatocellular carcinoma.
2. Must be 20 years of age or older.
3. Unresectable disease. Patients with resectable HCC but who refuse surgery may be enrolled after a documented consultation with a surgeon.
4. Radiologically measurable disease that is at least 2 cm in longest dimension of the target tumor.
5. ECOG performance status of ≤ 2.
6. Child-Pugh classification A.
7. Patients with chronic hepatitis B must be under long-term anti-viral agents with a high barrier of resistance, such as Entecavir, Tenofovir Disoproxil Fumarate, or Tenofovir Alafenamide.
8. Patients with chronic hepatitis C must reach sustained viral response by the treatment with any direct acting agent.
9. Acceptable hematologic, renal and liver function as follows within 28 days before entering the trial:

   (A)Absolute neutrophil count ≥ 1500/mm3 (B)Platelets ≥ 80,000/mm3 (C)Hemoglobin > 10.0 g/dL (D)Creatinine ≤ 2.0 mg/dl (E)Total bilirubin ≤ 1.5 mg/dl, unless due to Gilbert's syndrome (F)Transaminases (AST and ALT) ≤ 2 times above the upper limits (G)INR < 1.5
10. Patients must be able to provide informed consent.
11. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.
12. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Contraception must be continued for at least 5 months following the last dose of Nivolumab. Women of childbearing potential must have a negative pregnancy test. Women who have been menopausal for more than 1 year (more than 12 months since their last menstrual period) or patients who have undergone sterilization are not required to undergo pregnancy testing.

Exclusion Criteria:

1. Patients may not be receiving any other investigational agents, biological agents or other anti-cancer medication.
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring antibiotics (exception is a brief (≤10days) course of antibiotics to be completed before initiation of treatment), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Based on its mechanism of action and data from animal studies, Nivolumab can cause fetal harm when administered to a pregnant woman. Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
4. Has a diagnosis of primary immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
5. Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
6. HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <200 CD4+ T cells/microliter in the peripheral blood.
7. History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
8. Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps)
9. The target tumor is blocked by the bile duct or important blood vessel that leads to difficulty in intratumor injection.
10. Principal investigator believes that for one or multiple reasons the patient will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the patient.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve(ACU 0-22 weeks) | prior to the initial dose on day 1 and Day 3 of weeks 10, 14, 18 and 22.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve(ACU 0-24 weeks) | prior to the initial dose on day 2 of weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24.

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Zhongzheng Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No